CLINICAL TRIAL: NCT03612206
Title: Effect of Early Enteral Nutrition on Serum Acetylcholine Level and Inflammation in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Research Assistant, Nanjing PLA General Hospital
Other Study IDs: 2016NLYZDRC022
Record Dates: First submitted 2018-07-18; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Critical Illness; Enteral Nutrition; Inflammation
MeSH Terms: conditions — Critical Illness; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early enteral nutrition(EEN) is an important treatment for critical ill patients and attenuate systemic inflammation, but the mechanisms are not clear. Thus the investigator conducted this study to observe if EEN affects systemic inflammation though regulation of blood acetylcholine

ELIGIBILITY:
Inclusion Criteria:

* initiating enteral nutrition within the first 24-48h after intensive care unit (ICU) admission
* age more than 18 years
* Acute Physiology and Chronic Health Evaluation II (APACHE II) score >8

Exclusion Criteria:

* not expected to survive 24 hours
* pregnancy
* any terminal stage disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population mainly includes patients who suffered severe complications after surgery or severe trauma
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 14 months
  The number of survival and non-survival patients 28 days after inclusion
Intestinal barrier function within one week | 14 months
  The measurement of serum d-lactate was applied to evaluate the intestinal barrier function

REFERENCES:
- [Derived] Tao G, Min-Hua C, Feng-Chan X, Yan C, Ting S, Wei-Qin L, Wen-Kui Y. Changes of plasma acetylcholine and inflammatory markers in critically ill patients during early enteral nutrition: A prospective observational study. J Crit Care. 2019 Aug;52:219-226. doi: 10.1016/j.jcrc.2019.05.008. Epub 2019 May 10. PMID 31108325